CLINICAL TRIAL: NCT02170662
Title: Topical Bimatoprost Effect on Androgen Dependent Hair Follicles
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00017573
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-07

CONDITIONS: Male Pattern Hair Loss; Androgenetic Alopecia
Keywords: male pattern hair loss; androgenetic alopecia; bimatoprost
MeSH Terms: conditions — Alopecia | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active drug (Active Comparator): During Part I of the study, subjects will be randomized in a blinded fashion to either placebo (vehicle that does not contain active drug) or topical bimatoprost to apply to the scalp target area every day for 16 weeks. After a 10 day washout period, each group will be crossed over to the alternate topical preparation (Part II) to apply for 16 weeks.
  Interventions: Drug: Bimatoprost; Drug: Placebo
- Placebo (Active Comparator): During Part I of the study, subjects will be randomized in a blinded fashion to either placebo (vehicle that does not contain active drug) or topical bimatoprost to apply to the scalp target area every day for 16 weeks. After a 10 day washout period, each group will be crossed over to the alternate topical preparation (Part II) to apply for 16 weeks.
  Interventions: Drug: Bimatoprost; Drug: Placebo

INTERVENTIONS:
Drug: Bimatoprost — Bimatoprost 0.03% ophthalmic solution as purchased from the manufacturer will be the active drug.
Drug: Placebo

SUMMARY:
The purpose of this study is to determine the effect of bimatoprost solution on scalp hair growth. Bimatoprost 0.03% ophthalmic solution is currently approved by the FDA for treatment of glaucoma (Lumigan™) and for thickening of thin eyelashes (Latisse™). Bimatoprost 0.03% is not approved for the treatment of scalp hair loss and its use in this study is considered investigational which means it is still being tested in research studies.

Thirty-three subjects were consented and screened, 9 entered and 9 completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. Hamilton-Norwood patterns of baldness IIIV, IV, V, or VA.
2. Subject's hair color must have adequate contrast against scalp color to allow hair counting on macrophotography.
3. Good health with normal blood tests for hematological, renal, and liver function.
4. Able to return to Duke for study visits.

Exclusion Criteria:

1. ECOG >1.
2. Used topical or oral minoxidil in the past 6 months, oral finasteride in the past 12 months or oral dutasteride in the past 24 months.
3. Taken any warfarin, heparin, or retinoid for greater than 2 weeks during the past 6 months and any in the past month.
4. Taken any chemotherapy in the past 2 years.
5. Used any over-the-counter (OTC) preparation that purports to help hair growth in the past four months.
6. Used prostaglandins of any type in the past or currently.
7. Any history of alopecia areata, cicatricial alopecia, radiation to the head, hair transplants, or scalp reductions.
8. Any skin abnormalities in the target area that would effect hair growth.
9. Any history of glaucoma or elevated intraocular pressure (IOP).
10. Any cancer other than non-melanoma skin cancer (NMSC) in the past 2 years and all must be in remission.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise Olsen, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Bimatoprost: Part 1: Patients initially were randomized to apply placebo topically for 16 weeks.
  Between Part 1 and Part 2 subjects completed a 10 day washout period.
  Part 2: Patients were then randomized to apply active drug ( Bimatoprost 0.03% ophthalmic solution) topically for 16 weeks.
- Bimatoprost Then Placebo: Part 1: Patients initially were randomized to apply active drug ( Bimatoprost 0.03% ophthalmic solution) topically for 16 weeks.
  Between Part 1 and Part 2 subjects completed a 10 day washout period.
  Part 2: Patients were randomized to apply placebo topically for 16 weeks.
Period: Overall Study
Arm/Group | Placebo Then Bimatoprost | Bimatoprost Then Placebo
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Bimatoprost | Bimatoprost Then Placebo | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Target Area Total Hair Count
Description: The primary endpoint is the percent change in total hair count from the beginning and end of each part of the study.
Time Frame: Baseline to week 17; and week 17 to week 34
Population: intention to treat (ITT)
Measure: Mean (Full Range); unit: percentage change in total hair count
Arm/Group | Placebo Then Bimatoprost | Bimatoprost Then Placebo
Number analyzed (Participants) | 3 | 6
percentage change in total hair count
  Part 1: Baseline to week 17 | -2.6 [-10.4 to 2.7] | 27.4 [-19.8 to 112.5]
  Part 2: week 17 to week 34 | 4.9 [-2.4 to 12.0] | -5.8 [-33.3 to 10.4]

2. Secondary Outcome: Percent Change in the Target Area Terminal Hair Count
Description: Terminal hairs are those which grow beyond a cm and contribute to overall hair density.
Time Frame: Baseline to week 17; and week 17 to week 34
Measure: Mean (Full Range); unit: percent change of terminal hair count
Arm/Group | Placebo Then Bimatoprost | Bimatoprost Then Placebo
Number analyzed (Participants) | 3 | 6
percent change of terminal hair count
  Part 1: Baseline to week 17 | -2.1 [-9.8 to 10.1] | 12.1 [-18.7 to 32.5]
  Part 2: week 17 to week 34 | -5.1 [-22.7 to 8.2] | -8.3 [-25.0 to 14.1]

3. Secondary Outcome: Percent Change in the Target Area Vellus Hair Count
Description: Vellus hairs are fine hairs that generally do not grow beyond 1 cm and do not contribute to overall hair density. For the most part, they have a diameter of <40 um. They are increased in number in male pattern baldness
Time Frame: Baseline to week 17; and week 17 to week 34
Measure: Mean (Full Range); unit: Percent change of vellus hair count
Arm/Group | Placebo Then Bimatoprost | Bimatoprost Then Placebo
Number analyzed (Participants) | 3 | 6
Percent change of vellus hair count
  Part 1: Baseline to week 17; | -2.6 [-16.7 to 17.6] | 78.1 [-45.9 to 406.0]
  Part 2: week 17 to week 34 | 5.1 [-10.0 to 19.3] | 2.9 [-43.3 to 34.0]

4. Secondary Outcome: Percent Change in Hair Diameter
Description: The percent change in hair diameter is a recent addition to the methods of assessing efficacy of hair growth promoters. It is a measure of hair mass and does not separate out the effect on terminal and vellus hairs but rather combines the effect on both. Since it is only terminal hairs that contributes to normal hair density, this measure does not add anything to the measures of total, terminal and vellus hair counts in terms of overall effect on hair growth and is therefore not analyzed or reported here.
Time Frame: Baseline to week 17; Week 17 to week 34
Population: Data not analyzed, and therefore not reported.
Arm/Group | Placebo Then Bimatoprost | Bimatoprost Then Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo Then Bimatoprost | Bimatoprost Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes